CLINICAL TRIAL: NCT02865603
Title: Effectiveness of a Universal Classroom-based Preventive Intervention (PAX GBG) in Estonia: A Matched-pair Cluster-randomized Controlled Trial
Brief Title: Impact of PAX Good Behavior Game on Elementary School Students in Estonia
Acronym: PAXGBGEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Health Development, Estonia (Other Government)
Collaborators: European Social Fund (Other); Ministry of the Interior, Estonia (Unknown)
Responsible Party: Principal Investigator, Karin Streimann, Principal Investigator, National Institute for Health Development, Estonia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: T90-C305
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Mental Health Wellness 1; Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PAX Good Behavior Game (Experimental): The intervention is delivered by teachers within the normal school curriculum. Teachers from intervention classes completed 3-day training and were supported by the mentor, who visited their class during the 2016/17 school year and provided counseling via e-mail and phone. During the second year (2017/18) teachers could use the PAX GBG methods, but they did not receive additional support from the mentors.
  Interventions: Behavioral: PAX Good Behavior Game
- Waitlist control group (No Intervention): Control group continue their normal activities without intervention. After a post-test assessment in spring 2018 the control group teachers will be trained and supported to implement PAX GBG.

INTERVENTIONS:
Behavioral: PAX Good Behavior Game — PAX GBG includes evidence-based kernels and a classroom game where students are reinforced for their mutual success in withholding inappropriate behavior.
  Arms: PAX Good Behavior Game

SUMMARY:
The aim of this study is to measure the impact of the intervention (PAX GBG) in Estonian-language 1st grade classrooms on students' mental health and behaviour, and teacher's self-efficacy.

DETAILED DESCRIPTION:
2-year, matched-pair, cluster-randomized controlled trial with a intervention and wait-list control arm is conducted during school years 2016/17 and 2017/18. 42 volunteering schools were matched to pairs. One school in each pair was randomly selected to receive the PAX GBG or continue their normal activities without intervention. After a post-test assessment in spring 2018 the control group teachers are trained and supported to implement PAX GBG.

ELIGIBILITY:
Inclusion Criteria:

All schools with first grade classrooms and Estonian-language as instruction language in Estonia were qualified to take part of the study if they did fit the inclusion criteria.

Schools were suitable to participate if they:

* Had equal to or more than 13 pupils in the first grade classroom in 2016/17 school term;
* Did not implement any other evidence-based program in basic school stage 1 (grades 1-3), (for example KiVa bullying prevention program);
* Did not already implement PAX GBG;
* Had at least one first grade teacher who volunteers to participate for the whole study period of two years.

Exclusion Criteria:

* Schools for children with special educational needs and schools with Russian language as instruction language were excluded.
* Schools with single-sex classrooms were excluded.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 708 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in children's social and emotional well-being | Baseline, 7 months post-baseline and 19 months post-baseline
  Children's social and emotional well-being will be measured by the teacher-completed Strengths and Difficulties Questionnaire with impact supplement (SDQ; Goodman, 1999) and parent-rated Strengths and Difficulties Questionnaire (Goodman, 1997).

SECONDARY OUTCOMES:
Change in symptoms of attention deficit hyperactivity disorder (ADHD) among the children | Baseline, 7 months post-baseline and 19 months post-baseline
  The Swanson, Nolan and Pelham-IV Questionnaire (SNAP-IV) (Swanson et al., 2001) is an 18-item instrument for rating ADHD-related symptoms and will be completed by parents.
Change in children's behavioral inhibition | Baseline, 7 months post-baseline
  The effects of the intervention on inhibitory control will be measured using cognitive task (Go/No-Go task). The task will be developed specially for this research and completed by children.
Change in teachers' sense of efficacy | Baseline, 7 months post-baseline and 19 months post-baseline
  Teachers' efficacy will be measured with The Teachers' Sense of Efficacy Scale (TSES; Tschannen-Moran & Hoy, 2001). It is a self-reported measure for teachers that consists of 24 items and assesses the teacher's perception of their sense of effectiveness as a teacher.
Change in classroom behavior | Baseline, 7 months post-baseline and 19 months post-baseline
  Teacher-rated 4-item measure will be used to assess classroom behavior. The measure originates from Organisation for Economic Co-operation and Development (OECD) Teaching and Learning International Survey (TALIS) 2013 teacher's questionnaire (question nr 41) and asks to indicate how strongly does the teacher agree or disagree with statements about the classroom behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Streimann, Principal Investigator — National Institute for Health Development

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Streimann K, Selart A, Trummal A. Effectiveness of a Universal, Classroom-Based Preventive Intervention (PAX GBG) in Estonia: a Cluster-Randomized Controlled Trial. Prev Sci. 2020 Feb;21(2):234-244. doi: 10.1007/s11121-019-01050-0. PMID 31432379
- [Derived] Streimann K, Trummal A, Klandorf K, Akkermann K, Sisask M, Toros K, Selart A. Effectiveness of a universal classroom-based preventive intervention (PAX GBG): A research protocol for a matched-pair cluster-randomized controlled trial. Contemp Clin Trials Commun. 2017 Aug 30;8:75-84. doi: 10.1016/j.conctc.2017.08.013. eCollection 2017 Dec. PMID 29696198
- See also: PAX GBG Estonian web page — http://www.terviseinfo.ee/vepa